CLINICAL TRIAL: NCT05496868
Title: Phase 2, Randomized, Double-blinded, Placebo-controlled, Multicenter Study to Assess Efficacy and Safety of Reparixin as add-on Therapy to SoC in Acute Respiratory Distress Syndrome (RESPIRATIO)
Brief Title: Add-on Reparixin in Adult Patients With ARDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REP0122; 2022-001612-25 (EudraCT Number)
Record Dates: First submitted 2022-08-04; First posted 2022-08-11 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Acute Respiratory Distress Syndrome, Adult
Keywords: ARDS; Reparixin
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — reparixin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: the identity of the treatments will remain unknown to the subject, Investigator, site staff, CRO and Dompé's personnel until the study completion and formal unmasking. Only the Data Monitoring Committee (DMC) will have access to group-unblinded and/or fully unblinded DMC reports.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Reparixin + Standard of care (Experimental): Reparixin tablets 1200 mg TID (2 tablets x 600 mg TID) as add-on to the standard of care (SoC).
  Interventions: Drug: Reparixin 600mg
- Placebo + Standard of care (Placebo Comparator): Placebo tablets with the same schedule of reparixin, as add-on to the standard of care (SoC)
  Interventions: Other: Matching Placebo

INTERVENTIONS:
Drug: Reparixin 600mg — Reparixin 600 mg tablets, administered crushed through nasogastric tube at the dose of 1200 mg TID (2 tablets TID administered approximately about every 8 hours) as add-on to the standard of care. After extubation and if the patient can swallow, reparixin may be administered orally. Total duration of the treatment: 14 days
  Other Names: REP
  Arms: Reparixin + Standard of care
Other: Matching Placebo — Placebo tablets. Administered crushed through nasogastric tube with the same schedule as reparixin as add-on to the standard of care. After extubation and if the patient can swallow placebo may be administered orally.
  Total duration of the treatment: 14 days
  Other Names: Control
  Arms: Placebo + Standard of care

SUMMARY:
Study objectives

1. To characterize the efficacy of reparixin in ameliorating lung injury and systemic inflammation and expediting clinical recovery and liberation from mechanical ventilation in adult patients with moderate to severe ARDS (PaO2/FIO2 ratio ≤ 200).
2. to assess the effect of reparixin on systemic biomarkers linked to a hyper-inflammatory ARDS phenotype.
3. To evaluate the safety of reparixin vs. placebo in patients enrolled in the study.

DETAILED DESCRIPTION:
Phase 2, randomized, double-blinded, placebo controlled, multicenter study. All patients will receive therapy in line with current standard-of-care as it pertains to ARDS management (protocolized ventilator management will be made available to all sites in accordance with currently accepted standard of care). Patients will be randomized (1:1) to either reparixin or placebo. Duration of treatment will be 14 days. In this study the IMP will be either reparixin or matched placebo, which will be provided in the form of tablets to be disintegrated for naso-gastric tube administration or administered orally after extubation and between extubation and day 14 should the patient be able to swallow. In such cases the IMP may be administered either intact or crushed and mixed with a vehicle as per speech swallow evaluation.

The study will consist of 4 study periods:

Screening Randomization and Baseline assessments, Treatment (14 days with discretionary extension up to 21 days), Follow-up (up to 28 days or hospital discharge, whichever occurs first, and then up to day-60).

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent, according to local guidelines and regulation.
2. Male and female adults (>18 years old).
3. Mechanically ventilated (invasive) patients with PaO2/FIO2 ratio ≤200 in the presence of PEEP of ≥5 cmH20.
4. Respiratory failure not fully explained by cardiac failure or fluid overload (if acute Congestive Heart Failure exacerbation is identified as part of the clinical picture this should be addressed effectively and as soon as possible before the patient can be enrolled).
5. Bilateral radiologic opacities consistent with pulmonary edema on the frontal chest x-ray (CXR), or bilateral ground glass opacities on a chest computerized tomography (CT) scan.
6. ≤48 hours from fulfilling above ARDS criteria (if a patient is transferred from a non-participating hospital to a participating site a 12-hour period beyond the 48 hours is allowed)
7. Females of child-bearing potential who are sexually active must be willing not to get pregnant within 30 days after the last Investigational Medicinal Product (IMP) dose and must agree to at least one of the following reliable methods of contraception:

   1. Hormonal contraception, systemic, implantable, transdermal, or injectable contraceptives from at least 2 months before the screening visit until 30 days after the last IMP dose;
   2. A sterile sexual partner;
   3. Abstinence. In patients non able to personally consent to above due to complications of acute illness and/or its treatment assurances for the above must be given by LR and reiterated by patient when/if she is able to do so.

Female participants of non-child-bearing potential or in post- menopausal status for at least 1 year will be admitted. For all female subjects with child-bearing potential, pregnancy test result must be negative before first drug intake.

Exclusion Criteria:

1. Moderate-Severe chronic hepatic disease (as verified by a previously known Child-Pugh score ≥7). If baseline Child-Pugh score is not known it should not be calculated while the patient is acutely ill. In that case the patient is excluded on the basis of: ALT/AST ≥ 3x ULN and total bilirubin > 2x ULN or ALT/AST ≥ 5x ULN
2. Severe chronic renal dysfunction: eGFR (2021 CKD-EPI) < 30 mL/min/1.73m2. If baseline (chronic) renal function is not known the patient is only excluded if in need of acute renal replacement therapy (currently on RRT or to be imminently placed on RRT)
3. Participation in another interventional clinical trial.
4. Patients that are clinically determined to have a high likelihood of death within the next 24 hours based on PI's estimation.
5. Currently receiving ECMO or high frequency oscillatory ventilation.
6. Anticipated extubation within 24 hours of screening. (In such cases re-screening is allowed if the patient is within the enrollment window).
7. Evidence of GI dysmotility as demonstrated by presence of all the following: persistent gastric distention and enteral feeding intolerability and persistent gastric residuals >500 ml).
8. Anticipated transfer to a hospital not participating in the trial within 72 hours of screening.
9. Decision to withhold or withdraw life-sustaining treatment (patients may still be eligible however if they are committed to full support except cardiopulmonary resuscitation if cardiac arrest occurs).
10. History of:

    1. Documented allergy/hypersensitivity to sulfonamides, ibuprofen and other COX-1 and 2 inhibitors, and to the study product and/or its excipients.
    2. Lactase deficiency, galactosemia or glucose-galactose malabsorption.
    3. History of peptic ulcer, GI bleeding or perforation due to previous NSAID therapy.
11. Active bleeding (excluding menses) from uncontrolled site that cannot be definitively resolved prior to enrollment.
12. Pregnant or lactating women.
13. Women of childbearing potential and fertile men who do not agree to use at least one primary form of contraception during the study and up to 30 days after the last IMP dose. For patients non able to personally consent to above due to complications of acute illness and/or its treatment assurances for the above must be given by LR and reiterated by patient when/if he/she is able to do so.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
Change in oxygenation index (OI) from baseline to day 7 of treatment | to day 7
  The OI is defined as: % mean airway pressure x FIO2/PaO2
Ventilator free days (VFD) at day 28 | at day 28
  Number of days from successfully weaning to day 28; patients who died before weaning have no ventilator-free days

SECONDARY OUTCOMES:
Change in oxigenation index (OI) from baseline to day 4 | to day 4
  The lower the OI the better the outcome
Acute lung injury score at 2, 3, 7, 14 days (if still intubated) | at days 2, 3, 7, 14 (if still intubated)
  composite of PaO2/FIO2 ratio, PEEP, lung compliance (plateau airway pressure minus PEEP/TV) and extent of pulmonary infiltrates
Sequential Organ Failure Assessment (SOFA) score at 2, 3, 7, 14 days | at Days 2, 3, 7, 14 days (if still intubated)
Ventilatory ratio at 2, 3, 7, 14 days | at days 2, 3, 7, 14 days (if still intubated)
  product of minute ventilation and PaCO2
Incidence of Extracorporeal Membrane Oxygenation (ECMO) by day 14 | At day 14
Use of vasoactive medications by day 14 | At day 14
Chest X-Rays assessment of pulmonary edema by "radiographic assessment of lung edema" (RALE) score at 2, 3, 7, 14 days | at days 2, 3, 7, 14
Percentage of patients achieving pressure support ventilation equal to 5 cmH20 with PEEP equal to 5 cmH20 for 2 hours (measure of weaning) by day 28 and at hospital discharge | by day 28
Intensive Care Unit free days by day 28 and at hospital discharge | by day 28
Hospital-free days by day 28 and at hospital discharge | by day 28
Incidence of tracheostomies by day 28 and at hospital discharge | by day 28
Incidence of transfer to long term acute care (LTAC) facility by day 28 and at hospital discharge | by day 28
All-cause mortality by day 28 and 60 | by days 28 and 60
Change from baseline to day 3, 7 and 14 days in plasma levels of IL-6, IL-8, PAI-1, TNFr-1, ICAM-1 RAGE | Days 3, 7 and 14
Hospital discharge by day 28 | by day 28
Incidence of Treatment Emergent AEs (TEAEs) and SAEs (TESAEs) from the beginning of study treatment to up to the end of study participation. | from the date of First Patient First Visit (FPFV) to the date of Last Patient Last Visit (LPLV)

CONTACTS AND LOCATIONS:
Overall Officials: Moerer Onnen, MD, Principal Investigator — Universitaetsmedizin Goettingen
Locations (40):
- United States (33):
  - The University of Alabama at Birmingham Hospital, Birmingham, Alabama
  - Banner - University Medical Center Phoenix, Phoenix, Arizona
  - University of Southern California, Los Angeles, California
  - University of California Irvine Health, Orange, California
  - Unversity of California Davis Medical Center, Sacramento, California
  - Denver Health, Denver, Colorado
  - University of South Florida, Tampa, Florida
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Methodist Hospitals of Northwest Indiana, Gary, Indiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Newton Wellesley Hospital, Newton, Massachusetts
  - Baystate Health, Springfield, Massachusetts
  - Detroit Medical Center, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - MyMichigan Medical Center Midland, Midland, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Jackson Pulmonary Associates, Jackson, Mississippi
  - University of Missouri Health Care, Columbia, Missouri
  - Hackensack Meridian Health, Hackensack, New Jersey
  - NYU Langone Brooklyn, Brooklyn, New York
  - New York University Langone Health, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Oklahoma Medical Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Baptist Hospitals of Southeast Texas, Beaumont, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Cardiovoyage, Denison, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Utah Hospitals & Clinics, Salt Lake City, Utah
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Germany (6):
  - Universitaetsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitaetsmedizin Goettingen, Göttingen, Lower Saxony
  - Herzzentrum Muenster, Münster, North Rhine-Westphalia
  - Universitaetsklinikum Leipzig, Leipzig, Saxony
  - Berufsgenossenschaftliche Kliniken Bergmannstrost, Halle, Saxony-Anhalt
  - University Hospital of Schleswig-Holstein, Kiel, Schleswig-Holstein
- Ospedale San Raffaele, Milan, Lombardy, Italy

REFERENCES:
- [Derived] Truwit JD, Fleming K, Nanchal RS. Empowering Respiratory Therapists to Restrict Nebulized 3% Saline and N-Acetylcysteine During Mechanical Ventilation. Respir Care. 2025 Aug;70(8):937-945. doi: 10.1089/respcare.12586. Epub 2025 Feb 24. PMID 40028879

DOCUMENTS (2):
  • Study Protocol (2024-02-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT05496868/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-29): https://cdn.clinicaltrials.gov/large-docs/68/NCT05496868/SAP_001.pdf